CLINICAL TRIAL: NCT02969551
Title: Detection of Airway Obstruction by Manometry in Different Sleep Stages and Comparing it to DISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 88/14
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Manometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sleep apnea, Manometry and possibly DISE: Sleep apnea Patients recieved manometry measures and those who were not considered for CPAP Therapy recieved Drug induced sleep endoscopy.
  Interventions: Device: Manometry and possibly DISE

INTERVENTIONS:
Device: Manometry and possibly DISE — A Manometry is performed on all patients. After it in some Patient DISE is followed

SUMMARY:
Patients with OSA receive manometry measurements with Apneagraph (AG) during one night of sleep. All patients are simultaneously evaluated with polysomnography. Patients who are not eligible for CPAP therapy are additionally studied with drug-induced sleep endoscopy (DISE). The frequency and obstructions patterns in different sleep stages are assessed. In addition obstruction patterns detected with AG are compared with DISE examination in the selected cases.

ELIGIBILITY:
Inclusion Criteria:

* Apnea-Hypopnea-Index (AHI) ≥ 5.

Exclusion Criteria:

* age <18 years;
* body mass index (BMI) of >35 kg/m2; active infection;
* previous oral, head, or neck surgery in the last 3 months; pregnancy; chronic use of alcohol (> 60g ethanol per day or > 150g ethanol per week) or sedatives; illicit drug use;
* chronic obstructive pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a diagnosed obstructive sleep apnea Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Detection of obstruction depending of sleep stage | 8

SECONDARY OUTCOMES:
Comparing the manometry findings to DISE | 1 Hour

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Heiser, MD, Study Chair — attending doctor in ENT
Locations (1):
- Klinik für Hals- Nasen- Ohrenheilkunde, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No